CLINICAL TRIAL: NCT03943875
Title: GARDASIL 9: 3 Dose vs. 2 Dose With Delayed 3rd Dose
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19-0058; RP190022 (Other Grant/Funding Number: Cancer Prevention & Research Institute of Texas)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Immunization; Efficacy; Human Papilloma Virus
Keywords: HPV vaccination; Gardasil 9; vaccine efficacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Vials submitted for assay will be de-identified and labeled only with the study ID number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Females, 3 dose standard (Active Comparator): Three doses of the 9-valent HPV vaccine to be administered to the comparison group (15-26 years of age) at 0, 2, and 6 months.
  Interventions: Biological: 9-valent HPV vaccine, 3 doses standard timing
- Females, 2 dose with delayed 3rd dose (Experimental): Two doses of the 9-valent HPV vaccine to be administered to the experimental group (15-26 years of age) at 0 and 6 months. Additional HPV vaccine dose will be offered after final blood draw at 12 months.
  Interventions: Biological: 9-valent HPV vaccine, 2 dose efficacy
- Males, 3 dose standard (Active Comparator): Three doses of the 9-valent HPV vaccine to be administered to the comparison group (15-26 years of age) at 0, 2, and 6 months.
  Interventions: Biological: 9-valent HPV vaccine, 3 doses standard timing
- Males, 2 dose with delayed 3rd dose (Experimental): Two doses of the 9-valent HPV vaccine to be administered to the experimental group (15-26 years of age) at 0 and 6 months. Additional HPV vaccine dose will be offered after final blood draw at 12 months.
  Interventions: Biological: 9-valent HPV vaccine, 2 dose efficacy

INTERVENTIONS:
Biological: 9-valent HPV vaccine, 2 dose efficacy — Evaluate the efficacy of 2 doses of the HPV vaccine across a 12 month period following the 1st dose among 15-26 year old males and females.
  Arms: Females, 2 dose with delayed 3rd dose; Males, 2 dose with delayed 3rd dose
Biological: 9-valent HPV vaccine, 3 doses standard timing — Will be comparison group for 2 dose efficacy group.
  Arms: Females, 3 dose standard; Males, 3 dose standard

SUMMARY:
We are evaluating whether 15-26 year old males and females need a 3rd dose of the human papillomavirus (HPV) vaccine, or whether 2 doses provide similar protection as 3 doses from the 9 types of HPV that it protects against.

DETAILED DESCRIPTION:
The investigators are studying an amended dosing regimen of an approved drug (Gardasil 9) in the population for which it is approved (vaccine is approved for ages 9-45 years and participants in this study will be 15-26 years of age.) The purpose of the study is to examine a delayed dosing schedule. The current recommendation is to administer the vaccine in 3 doses (administered at 0, 1-2 months and 6 months) to those 15-26 years of age but only 2 doses (0 and 6 months) if given at 9-14 years of age. The investigators will conduct a randomized study to determine if 2 doses will elicit an immune response similar to the standard 3 doses in those 15-26 years of age. Participants in the study group will receive 2 doses of Gardasil 9 at 0 and 6 months. Participants in the control group will receive 3 doses of Gardasil 9 at 0, 1-2 months and 6 months. All participants (Target Accrual n=512) will have 5 mLs of blood drawn at 0, 7, and 12 months. Following the 12 month blood draw, participants randomized to 2-doses will receive the 3rd dose. Potential participants will be recruited in the University of Texas Medical Branch (UTMB) clinics where providers have given the PI permission to directly contact patients. The investigators will also display signs and use email announcements at UTMB and other college campuses and will advertise the study online or by mail. The investigators will call UTMB patients if their provider gave permission to contact the patient, or if the patients gave prior consent to contact through the UTMB system. Potential participants (and their parents, if under 18 years of age) will be screened with inclusion/exclusion criteria. Eligible and interested parents and patients will sign informed written consent. Patients under 18 years of age will sign written assent. At the initial visit, eligible, consented participants will have their blood drawn, be randomized into either the study or control group, and receive a dose of the HPV vaccine. Participants will be re-screened against the inclusion/exclusion criteria at subsequent visits. All participants will receive compensation administered through a ClinCard following each of the 3 blood draws.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 15-26 years old.
2. Ability to give informed consent. All participants under 18 years of age must have the informed consent of a parent and must assent to participation.
3. Has not received any prior doses of the HPV vaccine. We will ask the patient and his/her parent (if <18) about prior vaccination and check the state registry (Immtrac), as well as the UTMB electronic medical record (if previously seen at UTMB), We will check with their primary care provider, if feasible, for patients who are not a previously established UTMB patient.
4. Identified source of funding for vaccine which may include Texas Vaccines for Children (VFC) program, Medicaid, the Children's Health Insurance Plan (CHIP), Texas Healthy Women program or other public or private health insurance.
5. Reliable telephone access.
6. Participant and parent/ guardian (if <18) can read and speak either English or Spanish.

Exclusion Criteria:

1. For females, currently pregnant or plans to become pregnant or donate eggs in next 12 months. Sexually active females must report that they use regular birth control. All female subjects will be required to take a urine pregnancy test before each Gardasil 9 dose, unless it can be verified that she gave birth within the last week. Any subjects with positive tests at the initial visit will be disqualified from the study and advised to seek prenatal care. If a subject is pregnant when her follow-up visit window closes, she will be removed from the study.
2. History of 6 or more lifetime sexual partners.
3. History of any immunodeficiencies (HIV+, chemotherapy treatment, status splenectomy) or autoimmune disorders (lupus, thyroid disorder, psoriasis).
4. History of bleeding or platelet disorders such as hemophilia.
5. Currently taking medication which can suppress immune function including systemic corticosteroids, radiation therapy, cyclophosphamide, azathioprine, methotrexate, cyclosporine, leflunomide, TNF-alpha antagonists, monoclonal antibody therapies, or intravenous immunoglobulin treatment.
6. Known allergies to any components of the vaccine, including aluminum, yeast or Benzonase.
7. Febrile at ≥100°F in the 24 hours prior to vaccination. This will be reviewed before each Gardasil 9 dose.
8. Received any non-study inactive vaccines within the past 14 days or any live vaccines within the past 30 days. Those excluded for this reason will be re-screened under the same study number at a later date.
9. Plan to move out of the Galveston/Houston area in the 13 months following study entry.

Ages: 15 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 757 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Short-term human papillomavirus (HPV) type-specific antibody response for type HPV-6 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 6, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-11 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 11, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-16 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 16, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-18 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 18, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-31 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 31, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-33 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 33, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-45 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 45, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-52 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 52, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-58 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (no detectable antibodies) to seropositive (antibodies at or exceeding natural immunity levels) to HPV type 58, measured as number of participants.
HPV type-specific antibody response for type HPV-6 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 6. Measured as number of participants.
HPV type-specific antibody response for type HPV-11 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 11. Measured as number of participants.
HPV type-specific antibody response for type HPV-16 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 16. Measured as number of participants.
HPV type-specific antibody response for type HPV-18 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 18. Measured as number of participants.
HPV type-specific antibody response for type HPV-31 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 31. Measured as number of participants.
HPV type-specific antibody response for type HPV-33 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 33. Measured as number of participants.
HPV type-specific antibody response for type HPV-45 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 45. Measured as number of participants.
HPV type-specific antibody response for type HPV-52 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 52. Measured as number of participants.
HPV type-specific antibody response for type HPV-58 | Month 12
  Yes/ No count, Number of patients with an antibody level at or above predetermined cutoff (natural immunity) for HPV type 58. Measured as number of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Abbey B Berenson, MD, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Berenson AB, Panicker G, Unger ER, Rupp RE, Kuo YF. Immunogenicity of 2 or 3 Doses of 9vHPV Vaccine in U.S. Female Individuals 15 to 26 Years of Age. NEJM Evid. 2024 Feb;3(2):EVIDoa2300194. doi: 10.1056/EVIDoa2300194. Epub 2024 Jan 23. PMID 38320488